CLINICAL TRIAL: NCT03459001
Title: A Prospective, Observational Study to Evaluate the Use of a High Calorie, High Protein Tube Feeding Product in an Adult Population With or at Risk of Malnutrition
Brief Title: Evaluation of a High Calorie, High Protein Tube Feeding Product in an Adult Population With or at Risk of Malnutrition
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: BL32
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tube Fed Malnourished Outpatients: Outpatients that are malnourished or at risk of malnutrition and have been placed on a nutritional care plan, which includes a complete tube feeding formula as sole source nutrition
  Interventions: Other: Tube Feeding Product

INTERVENTIONS:
Other: Tube Feeding Product — a high calorie, high protein tube feed product consumed sole source per their physician's recommendation and per standard of care

SUMMARY:
This prospective, observational study is designed to observe the use of a high calorie, high protein tube feed product in adults that are malnourished or at risk of malnutrition, as assessed by a clinician, and have been placed on a nutritional care plan which includes a tube feeding formula, per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Malnourished or at risk for malnutrition based on the Malnutrition Universal Tool (MUST) score ≥ 2.
* Under the care of a health care professional for malnutrition or at risk of malnutrition and has been prescribed the study formula.
* Requires and agrees to be tube fed the enteral feeding product for at least 16 consecutive days as their sole-source of nutritional intake.
* Free living in the community or is residing in a nursing home.
* Conforms to the requirements set forth on the study product label.

Exclusion Criteria:

* Currently taking or has taken antibiotics within 2 weeks prior to enrollment.
* Consuming food PO.
* Current active cancer and the study physician determines that the subject is not suitable for the study.
* History of diabetes mellitus as evidenced by taking anti-hyperglycemic medications or by self-reported dietary modification for control of diabetes mellitus.
* Renal or liver failure.
* Pregnant as demonstrated by self-report.
* Severe auto immune disease (per physician's discretion) and is on immuno-modulating therapy.
* History of allergy to any of the ingredients in the study product.
* Active Human Immunodeficiency Virus (HIV).
* Known dementia, brain metastases, eating disorders, history of significant neurological or psychiatric disorder, or any other psychological condition that may interfere with study product consumption and does not have a caregiver who can assist them with adherence to the study protocol.
* Condition that is contraindicated to tube feeding the study product.
* Taking part in a non-approved clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients ≥ 18 years of age that are malnourished or at risk of malnutrition and have been placed on a nutritional care plan, which includes a complete tube feeding formula as sole source nutrition will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Tube Feed Product Compliance | Day 1 to Day 20
  Average Daily Intake and Proportion of Days Compliant

SECONDARY OUTCOMES:
Adverse Events | Day 0 to Day 20
  Non serious AE and SAE collection
Body Mass Index | Day 0 to Day 20
  Weight, Height

CONTACTS AND LOCATIONS:
Overall Officials: Maria Camprubi Robles, PhD, Study Chair — Abbott Nutrition
Locations (9):
- Spain (9):
  - Residencia Plata y Castañar, Madrid
  - Residencia Albertia Moratalaz, Madrid
  - Residencia Valle de la Oliva, Madrid
  - Hospital Clinico de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital La Fe 3065, Valencia
  - Hospital La Fe 3066, Valencia
  - Hospital La Fe de Valencia 3033, Valencia
  - Hospital La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided